CLINICAL TRIAL: NCT03689738
Title: Effects of Potato Resistant Starch Intake on Insulin Sensitivity, Related Metabolic Markers and Satiety in Men and Women at Risk for Type 2 Diabetes
Brief Title: Effects of Potato Resistant Starch Intake on Insulin Sensitivity, Related Metabolic Markers and Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Alliance for Potato Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: MB-1802
Record Dates: First submitted 2018-09-27; First posted 2018-09-28 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Insulin Sensitivity; Lipid Metabolism; Resistant Starch; Potato
Keywords: Resistant Starch; Free Fatty Acids; Potato; Insulin sensitivity; Lipid Metabolism
MeSH Terms: conditions — Insulin Resistance | interventions — Resistant Starch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Potato condition (Experimental): Potato lunch and dinner meals, and an evening snack containing 100 g potatoes and 5 g RS per meal, providing a total of 300 g/d potatoes, equivalent to roughly two whole potatoes, and 15 g/d RS.
  Interventions: Other: Potato (Resistant Starch)
- Control condition (Active Comparator): Isocaloric, CHO-matched, low-fiber, RS-free lunch and dinner meals, and an evening snack.
  Interventions: Other: CHO-matched (Low-fiber, RS-free)

INTERVENTIONS:
Other: Potato (Resistant Starch) — Potato lunch and dinner meals, and an evening snack containing 100 g potatoes and 5 g resistant starch (RS) per meal, providing a total of 300 g/d potatoes, equivalent to roughly two whole potatoes, and 15 g/d RS.
  Arms: Potato condition
Other: CHO-matched (Low-fiber, RS-free) — Isocaloric, CHO-matched, low-fiber, RS-free lunch and dinner meals, and an evening snack.
  Arms: Control condition

SUMMARY:
The objective of this study is to assess whether intake of baked and then chilled potatoes over a 24-h period, compared to intake of isocaloric, carbohydrate (CHO)-matched foods low in fiber and resistant starch (RS), will increase insulin sensitivity, breath hydrogen and satiety, and decrease hunger and free fatty acid (FFA) levels in overweight or obese men and women at risk for metabolic syndrome and diabetes mellitus.

DETAILED DESCRIPTION:
This randomized, two-period crossover study will include one screening/baseline visit (visit 1) and two 24-h treatment periods (treatment period 1: visits 2 and 3 and treatment period 2: visits 4 and 5). A minimum 7-d washout will occur between the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a male or female, 18-74 years of age, inclusive.
2. Subject has a BMI of ≥27.0-39.99 kg/m2 at visit 1.
3. Subject has a waist circumference ≥40 in for men and ≥35 in for women at visit 1.
4. Subject has a rating of 7 to 10 on the Vein Access Scale at visit 1 (Appendix 2).
5. Subject is willing to maintain a stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial, except for the substitution of the study foods.
6. Subject is willing to consume the study foods provided throughout the duration of the study.
7. Subject has no plans to change smoking habits or other nicotine use during the study period and is willing to refrain from nicotine use for 1 h prior to and during all test visits.
8. Subject is willing to refrain from alcohol and vigorous physical activity 24 hours prior to test days (visits 2, 3, 4 and 5).
9. Subject is judged by the Investigator to be in general good health on the basis of medical history.
10. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has a fasting capillary glucose of ≥126 mg/dL and/or a HbA1C ≥6.5 % based on the capillary blood draw at visit 1.
2. Subject has a history or presence of atherosclerotic cardiovascular disease, chronic inflammatory disease (including irritable bowel disease, lupus, rheumatoid arthritis), or clinically important endocrine (including type 1 or type 2 diabetes mellitus), pulmonary (including uncontrolled asthma), hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric, or biliary disorders.
3. Subject has a history of cancer in the prior 5 years, except for non-melanoma skin cancer.
4. Subject has experienced a change in body weight of ±4.5 kg (10 lbs) over the 3 months prior to visit 1.
5. Subject has a known allergy, sensitivity, or intolerance to any ingredients in the study foods.
6. Subject has uncontrolled hypertension (systolic BP ≥160 mm Hg or diastolic BP

   * 100 mm Hg) at visit 1.
7. Subject has unstable use of any antihypertensive medication within 4 weeks prior to visit 1. Unstable use is defined as initiation or dose alteration.
8. Subject has used any of the following medications within 4 weeks of visit 1:

   1. With the exception of the stable use of statins (defined as no initiation or dose alteration within 4 weeks of visit 1) any medications intended to alter the lipid profile, including but not limited to: bile acid sequestrants, cholesterol absorption inhibitor, fibrates, niacin (drug form), omega-3-ethyl ester drugs, and/or proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors.
   2. Medications known to significantly influence carbohydrate metabolism, including, but not limited to, adrenergic receptor blockers, diuretics, and/or hypoglycemic medications.
   3. Weight-loss drugs (including over-the-counter medications) or weight loss programs.
   4. Systemic corticosteroid drugs.
9. Subject has used any of the following foods or dietary supplements within 2 weeks of visit 1:

   1. Food/supplements known to influence lipid metabolism, including, but not limited to, omega-3 fatty acid supplements (e.g., flaxseed, fish or algal oils) or fortified foods, sterol/stanol products; dietary supplements (red rice yeast supplements; garlic supplements; soy isoflavone supplements; niacin or its analogues at doses >400 mg/d (or others at the discretion of the Investigator).
   2. Irregular or inconsistent use of Metamucil® or other viscous fiber-containing supplements (consistent, daily use up to 1 tsp of a viscous-fiber supplement is acceptable).
10. Subject has used antibiotics within 5 days of any clinic visit: For those with an active infection and/or using antibiotics, subjects must wait at least 5 d after the infection resolves or antibiotic use is complete. The test period will be extended for study completion in these cases.
11. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
12. Subject has extreme dietary habits (e.g. very low CHO diet, vegan, etc.).
13. Subject has a history of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.
14. Subject is a habitual breakfast skipper (defined as skipping breakfast ≥4 times per week).
15. Subject has a current or recent history (past 12 months), or strong potential, for drug or alcohol abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1 ½ oz distilled spirits).
16. Subject has been exposed to any non-registered drug product within 30 days of visit 1.
17. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Change in the Matsuda insulin sensitivity index (MISI) | Up to 300 minutes - measured at the end of each treatment period
  Difference in the Matsuda insulin sensitivity index (MISI) between the Potato and Control conditions following a breakfast meal tolerance test (MTT) completed on day 2 of each treatment period.

SECONDARY OUTCOMES:
Change in the total area under the curve (AUC) for insulin | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the total area under the curve (AUC) from pre-breakfast intake to 5-h post-breakfast intake for insulin.
Change in the total area under the curve (AUC) for glucose | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the total area under the curve (AUC) from pre-breakfast intake to 5-h post-breakfast intake for glucose.
Change in the incremental AUC (iAUC) for insulin | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the incremental AUC (iAUC) from pre-breakfast intake to 5-h post-breakfast intake for insulin and glucose.
Change in the incremental AUC (iAUC) for glucose | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the incremental AUC (iAUC) from pre-breakfast intake to 5-h post-breakfast intake for insulin and glucose.
Change in the AUC for FFA | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the AUC for FFA from 0-3 h, 0-5 h, and 3-5 h postprandially.
Change in the net iAUC for fullness, hunger, desire to eat and prospective food consumption | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the net iAUC from pre-breakfast intake to 5-h post-breakfast intake for fullness, hunger, desire to eat and prospective food consumption.
Change in the total AUC for breath hydrogen | Up to 300 minutes - measured at the end of each treatment period
  Differences between the Potato and Control conditions following a breakfast MTT completed on day 2 of each treatment period in the total AUC for breath hydrogen from 0-5 h post-breakfast intake.

CONTACTS AND LOCATIONS:
Locations (1):
- Cathy Maki, Boca Raton, Florida, United States